CLINICAL TRIAL: NCT00214292
Title: A Pilot Study of Intraoperative Margin Assessment Comparing Optical Spectroscopy and Frozen Section Analysis for Ductal Carcinoma In Situ of the Breast
Brief Title: Evaluation of Breast Cancer Surgical Margins Using Optical Spectroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M-2002-0211; 2002-211 (Other: MR IRB)
Record Dates: First submitted 2005-09-14; First posted 2005-09-21 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Spectrometry, Fluorescence

INTERVENTIONS:
Procedure: fluorescence spectroscopy and diffuse spectroscopy

SUMMARY:
This study will apply optical spectroscopy to intraoperative margin assessment during surgery for breast cancer. We hypothesize that a combination of fluorescence spectroscopy and diffuse reflectance spectroscopy will reliably detect involved surgical margins. Twenty patients with ductal carcinoma in-situ will undergo a standard lumpectomy followed by scanning with a sterile optical spectroscopy probe. Frozen sections from the surgical cavity will be used to evaluate the margins. Optical spectroscopy data will be categorized as benign or malignant using a statistical algorithm and the results will be compared with the frozen and permanent section results.

ELIGIBILITY:
Inclusion Criteria:

* ductal carcinoma in-situ or invasive carcinoma diagnosed by image directed core biopsy who are planning to undergo breast conserving surgery

Exclusion Criteria:

* patients who were diagnosed with excisional biopsy and patients undergoing mastectomy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2005-05; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
The goal of this research is to develop a minimally invasive technology with the capability of rapidly assessing surgical margins for breast cancer patients undergoing breast conserving therapy.

SECONDARY OUTCOMES:
Two potential benefits from developing this technology are:
1. Decreasing operative times by eliminating the need to wait for histologic margin assessment.
2 Intraoperative margin assessment will become available for surgeons performing breast conserving therapy in facilities in-house pathologists.

CONTACTS AND LOCATIONS:
Overall Officials: Tara Breslin, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States